CLINICAL TRIAL: NCT05023122
Title: The Effect of Oral Vitamin D Supplements on Fusion Outcome in Patients Receiving Elective Lumbar Spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Show Chwan Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pei-Yuan Lee, MD, Honorary President, Show Chwan Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RD105014
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Vitamin D; Spinal Fusion; Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vitamin D3 + calcium (Experimental): vitamin D3 (cholecalciferol) 800 IU QD and calcium citrate 600 mg QD, given from postoperative day 1 and lasted for 3 months
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: calcium
- calcium only (Active Comparator): only calcium citrate 600 mg QD, given from postoperative day 1 and lasted for 3 months
  Interventions: Dietary Supplement: calcium

INTERVENTIONS:
Dietary Supplement: vitamin D3 — vitamin D3 (cholecalciferol) 800 IU QD
  Arms: vitamin D3 + calcium
Dietary Supplement: calcium — calcium citrate 600 mg QD

SUMMARY:
The process of bony fusion is a dynamic bone remodeling process and a variety of risk factors have been identified to contribute to pseudoarthrosis.Vitamin D deficiency has been reported to be associated with more pseudoarthrosis, prolonged time to fusion, and poorer spine function and quality of life after spinal fusion.However, as the review article presented, it lacks high-quality evidence to investigate the role of vitamin D supplements in spinal fusion. Therefore, this randomized controlled trial aimed to evaluate the effectiveness of oral vitamin D supplements on fusion outcomes in patients receiving elective lumbar spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 80 years
* Indicated of elective spine fusion surgery for spinal stenosis or degenerative spondylolisthesis at the study hospital from January 2016 to December 2017.

Exclusion Criteria:

* Spinal instability due to trauma, infection, or malignancy
* History of previous spine surgery
* Hemodialysis
* Long-term steroid use
* History of medical treatments for osteoporosis
* Postoperative follow-up for less than 12 months
* Newly-onset compression fracture after study procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
fusion rate at postoperative 1 year | postoperative 1 year
  Fusion status were assessed by radiography and computed tomography of the lumbar spine. Fusion was defined as the presence of bridging callus without radiolucent line, spinal range of motion between two fused vertebrae less than 5 degrees, and no implant loosening or failure on lumbar spine radiography.

SECONDARY OUTCOMES:
time to fusion | from postoperative day 1 to postoperative 1 year
  Time to fusion were assessed by radiography and computed tomography (CT) of the lumbar spine.Fusion was defined as the presence of bridging callus without radiolucent line, spinal range of motion between two fused vertebrae less than 5 degrees, and no implant loosening or failure on lumbar spine radiography
spine function at postoperative 3 months | postoperative 3 months
  Spine function was evaluated using Oswestry Disability Index (ODI), which contains 10 patient-completed questions addressing spinal function. Each question is presented as 6-point Likert scales from 0 to 5 (0 = best outcome, 5 = worst outcome). The overall ODI score ranges from 0% to 100% and a lower score indicates better function.
spine function at postoperative 6 months | postoperative 6 months
  Spine function was evaluated using Oswestry Disability Index (ODI), which contains 10 patient-completed questions addressing spinal function. Each question is presented as 6-point Likert scales from 0 to 5 (0 = best outcome, 5 = worst outcome). The overall ODI score ranges from 0% to 100% and a lower score indicates better function.
pain at postoperative 3 months | postoperative 3 months
  Degree of pain was evaluated using visual analogue scale (VAS), which ranges from 0 to 10 (0 = least pain, 10 = worst pain).
pain at postoperative 6 months | postoperative 6 months
  Degree of pain was evaluated using visual analogue scale (VAS), which ranges from 0 to 10 (0 = least pain, 10 = worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, PhD, Study Director — Show Chwan Memorial Hospital, Changhua, Taiwan
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu MH, Tseng YK, Chung YH, Wu NY, Li CH, Lee PY. The efficacy of oral vitamin D supplements on fusion outcome in patients receiving elective lumbar spinal fusion-a randomized control trial. BMC Musculoskelet Disord. 2022 Nov 18;23(1):996. doi: 10.1186/s12891-022-05948-9. PMID 36401234